CLINICAL TRIAL: NCT02097667
Title: EVERREST - Developing a Therapy for Fetal Growth Restriction. A 6 Year Prospective Study to Define the Clinical and Biological Characteristic of Pregnancies Affected by Severe Early Onset Fetal Growth Restriction.
Brief Title: EVERREST Developing a Therapy for Fetal Growth Restriction
Acronym: EVERREST
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Hospital Clinic of Barcelona (Other); Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 13/0289
Record Dates: First submitted 2013-10-31; First posted 2014-03-27 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Fetal Growth Retardation
Keywords: Severe early onset Fetal Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, whole blood, fixed placenta, frozen placenta, fixed placenta bed.
Oversight: Data Monitoring Committee: No

SUMMARY:
Fetal Growth Restriction (FGR) is a major obstetric problem, affecting 1.46 million fetuses worldwide each year and contributing to 50% of stillbirths. Severe early onset FGR affects 1 in 500 pregnancies, leading to stillbirth or the need for delivery before 28 weeks gestation. The combination of FGR and prematurity is associated with a significant risk of neonatal mortality and short and long-term complications. Even modest increases in birthweight (e.g from 500 to 600g) and gestation at delivery (e.g from 26 to 27 weeks) are associated with significantly better outcomes but there are currently no treatments.

The EVERREST Clinical Trial, funded by the European Commission, aims to develop a treatment which will increase fetal growth in severe early onset FGR. It will use gene therapy injected into the uterine arteries of the mother to increase the levels of vascular endothelial growth factor (VEGF) and so increase uterine artery blood flow and fetal growth.

The EVERREST prospective study aims to form a clinical database and biobank of pregnancies affected by severe early onset FGR to improve understanding of the condition and serve as a comparison to assess the safety and efficacy of this intervention.

The prospective study will take place across four European centers who will later take part in the EVERREST Clinical Trial. Women with singleton fetuses with early onset FGR will be approached to take part in the study. Participating women will provide blood samples, details of their clinical condition, samples of umbilical cord blood, placenta and myometrial and placental bed biopsies at the time of Caesarean section (if needed). Data on short and long-term outcomes of the babies will be collected. All data will be entered onto a central database for eventual use as a comparator for treated women on the EVERREST Clinical Trial, for which separate ethical approval will be sought.

DETAILED DESCRIPTION:
Fetal Growth Restriction (FGR) is a major obstetric problem, affecting 1.46 million fetuses worldwide each year and contributing to 50% of stillbirths. Severe early onset FGR affects 1 in 500 pregnancies, leading to stillbirth or the need for delivery before 28 weeks gestation. The EVERREST prospective study plans to clinically and biochemically characterise a cohort of pregnancies affected by severe early onset FGR across the four European centres. A database will be created containing information about antenatal investigations, maternal complications, fetal outcome and neonatal progress. This will be linked to a biobank containing samples of maternal blood, umbilical cord, umbilical cord blood, placenta, placental bed and myometrium.

There are three aims to this study:

1. To provide data from pregnancies affected by severe early onset FGR with which to compare outcomes from a group of pregnancies that will undergo treatment using maternal Ad.VEGF gene therapy.
2. To provide important information about the likely prognosis for babies born after affected pregnancies in the short and long term. These are data which are currently lacking.
3. To provide samples that will be used to investigate the biological mechanisms that underlie the condition, which subsequently may be used to provide biomarkers of outcome.

The design of the project has involved consultation with leading European fetal medicine specialists, neonatologists, pathologists and biomedical scientists who form part of the EVERREST consortium. The multicenter nature of the project raises issues of confidentiality and data protection but also allows for a larger data set from which to draw more meaningful conclusions. Furthermore it means that the findings are applicable not just in the United Kingdom but also in Europe. It also provides a larger group of patients from which to recruit to the EVERREST trial. The project has also been given approval by the National Institute for Health Research, funded Fetal Medicine Clinical Study Group at the Royal College of Obstetrician and Gynecologists, of which the PI is a member. Other leading Fetal Medicine centres across the United Kingdom will be involved in recruiting to the prospective study so that a wider picture of severe FGR and samples from affected pregnancies are available in the UK.

Recruitment Women referred to the Fetal Medicine Unit for suspected severe early onset Fetal Growth Restriction will be given a Participant Information Sheet (PIS) to read. If the diagnosis of severe early onset FGR is made women will be asked if they are interested in taking part in the study. Interested eligible women will meet with a member of the research team who will read through the PIS with them and answer any questions they have. If the woman would like more time to decide they can meet with a member of the research team at a subsequent hospital appointment.

Risks, burdens and benefits Women may be distressed by discussing the study at what will already be a worrying and upsetting time following the diagnosis of severe early onset FGR. If this is the case it will not be pursued, and can be discussed at a future appointment if the woman wishes. Within the University College London Hospital Fetal Medicine Unit women are frequently given information about research at the time of their appointments and the investigators have not found this to be distressing to them.

Women may be concerned that declining to be involved in the study will affect the care that they receive. The Participant Information Sheet will make it clear that this will not be the case.

There is a risk of breach of confidentiality with data sharing. This will be minimised by holding data in a central secure database, which will be password protected and can only be accessed by authorised members of the team, and by creating a unique pseudoanonymised Participant Identification Number which will be used on the database. Participant identifiable data, including name, address and hospital ID number, will not be entered onto the central database.

Performing the ultrasound assessments of uterine artery blood flow will add 2-5 minutes to a 30 minute ultrasound scan. At these appointments women will often need to wait for their ultrasound scan and may need blood pressure monitoring, urine checks and fetal heart beat monitoring (cardiotocograph) as part of their routine care. This can mean they are at the hospital for an hour or more, or which the uterine blood flow assessment would be a small fraction.

The maternal blood samples may involve temporary pain and/or bruising. This will be minimised by having the samples taken by trained healthcare professionals. During a low risk pregnancy two routine blood samples are recommended at booking and 28 weeks gestation. In pregnancies complicated by severe early onset FGR several additional blood samples will be needed as part of clinical care. Investigators plan to take the investigators first sample at the same time as blood tests needed to look for maternal infections (toxoplasmosis, cytomegalovirus, rubella) and the investigators second at the same time as pre-operative blood tests taken before Caesarean section.

The myometrial biopsy and placental bed biopsy will each add an estimated 1 minute to the Caesarean section. Generally the surgical time for a Caesarean is about 45 minutes but when anesthetic time and patient transfer are included the overall procedure takes approximately 2 hours. They are not associated with a significant risk of hemorrhage or post-operative complications. Biopsies would not be taken if there were a clinical contra-indication e.g. excessive uterine bleeding or maternal medical conditions meaning the duration of the surgery had to be limited.

The umbilical cord, umbilical cord blood and placental samples will be taken after the baby has been delivered, the cord cut and the placenta delivered so will not involve any pain or inconvenience for the mother or baby.

At the moment there is no treatment for severe early onset FGR. This can leave parents feeling helpless in the face of the diagnosis. It may help them to feel their participation could contribute to a better understanding of the condition and a potential treatment in the future. Women who have a pregnancy affected by severe early onset FGR are at higher risk of having a future affected pregnancy, so there may also be the potential for a direct benefit to their future reproductive health.

Babies born from pregnancies affected by severe early onset FGR are routinely followed up in all four EU countries to two years of age, corrected for prematurity, since it is well known that many have severe morbidity for which medical input is required. Investigators will collect data about clinical blood results, investigations and neurodevelopmental assessments, which are performed routinely as part of their standard care.

Confidentiality The EVERREST consortium will be collecting demographic and clinical data about participants from four European countries which will be combined in a central database.

Within each centre participants will be given a unique study Participant Identification Number (PIN). Data will be entered under this identification number onto the central database stored on the servers based at the University College London. The database will be password protected and only accessible to members of the EVERREST Consortium, UCL Clinical Trials Unit, the participating hospitals and external regulators, including the European Commission. The servers are protected by firewalls and are patched and maintained according to best practice. The physical location of the servers is protected by Closed-circuit television and security door access. The database and coding frames will be developed by the Trial Manager in conjunction with the CTU.

The information linking participant identifiable data to the pseudoanonymised Participant Identification Number will be held locally by the research sites. This will either be held in written form in a locked filing cabinet or electronically in password protected form on hospital computers. After completion of the study the data linking participant identifiable data to the PIN will be destroyed and the database will be retained on the servers of University College London for on-going analysis in conjunction with the bio bank.

All members of the research team will receive training in the regulations surrounding confidentiality and data handling and their responsibilities in this area. It will be made clear to participants in the PIS and during the process of consent that data will be obtained from their medical records and the medical records of their baby. It will be explained that this data will be stored in a form in which they are not directly identifiable and will be shared within the European Union for the purposes of the study. Electronic data will be transferred in encrypted and password protected form.

It is not anticipated that the results of analysing the tissue samples will have any direct clinical significance for the participants. If, however, results were to be obtained which would have a serious impact on the participant's current or future health these would be fed back to the recruiting study centre under the Participant Identification Number. Within the recruiting centre the results could be linked back to the participant without them being identified to the rest of the research team.

Use of tissue samples in future research At the conclusion of the study, stored samples will be transferred to a site with national regulatory approval, for retention as a bio bank. Participant consent will be obtained in advance for this retention. Separate ethical application will be made for research using these samples. Samples will be stored until they are fully used or become unusable, which is anticipated to be a maximum of 10 years for frozen samples.

If participants do not give their consent for retention for future research then UK samples will be disposed of in accordance with the Human Tissue Authority's Code of Practice and European samples will be disposed of according to local and national guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Live singleton fetus
* Estimated fetal weight <600g and <3rd centile for gestational age as defined by local criteria
* Gestational age at diagnosis 20+0-26+6 weeks, based on ultrasound and/or last menstrual period
* Informed consent given by the participant and signed consent form completed

Exclusion Criteria:

* Multiple pregnancy
* Maternal age under 18 years
* Known abnormal karyotype at enrolment
* Known structural abnormality at enrolment defined as a lethal, incurable serve abnormality with a high risk of residual handicap.
* Indication for immediate delivery
* Participants who lack the capacity to give informed consent
* Any medical or psychiatric condition which compromises the participant's ability to participate
* Maternal HIV or hepatitis B or C infection
* Premature preterm rupture of membranes before enrolment

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with FGR
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
data collection from pregnancies affected by severe early onset FGR. | each hospital visit and up to 2 years follow up for babies
  As the study will be purely descriptive there are no defined primary outcome measures. Data will be collected on the following:
  * Parental demographics
  * Maternal past medical history and obstetric history
  * Antenatal ultrasound findings including growth and Doppler measurements
  * Maternal antenatal, perinatal and postnatal complications and treatment
  * Stillbirth
  * Delivery and immediate neonatal condition
  * Neonatal progress including complications, treatment and neonatal death
  * Infant growth and development up to 2 years corrected age
  * Maternal and neonatal service use

OTHER OUTCOMES:
Model validation 1 | 2021
  The following models, developed in a discovery set of n=63, will be validated in the remaining participants. Model parameters are transformed values of maternal serum protein concentrations or normalised protein expression. Model estimates (area under the curve (AUC) and 95% confidence intervals (95%CI)) are from leave-one-out cross-validation for outcomes 1 and 2 and from 5-fold cross-validation with bootstrap bias CI correction for outcome 3.
  Outcome 1: fetal or neonatal death
  1. Placental growth factor (PlGF): AUC 0.749 (95%CI 0.615-0.883)
  2. PlGF & lymphotactin: AUC 0.839 (0.731-0.947)
  3. PlGF, lymphotactin & fibronectin: AUC 0.848 (0.735-0.961)
Model validation 2 | 2021
  Outcome 2: Fetal death or delivery <28+0 weeks of gestation
  1. PlGF: AUC 0.858 (0.760-0.956)
  2. PlGF & pregnancy specific beta-1 glycoprotein 1 (PSG1): AUC 0.906 (0.818-0.994)
  Outcome 3: Development of umbilical artery pulsatility index (UmAPI) >95th centile (Schaffer & Stauch) in pregnancies with UmAPI <95th centile at enrolment
  1. PlGF: AUC 0.844 (0.495-0.950)
  2. PlGF & fibronectin: AUC 0.900 (0.620-0.991)

CONTACTS AND LOCATIONS:
Overall Officials: Anna David, Dr, Principal Investigator — Institute of Women's Health, UCL
Locations (4):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Maternal-Fetal Unit Hospital Clinic de Barcelona, Barcelona, Spain
- Lund University Hospital and University Hospital Malmö, Malmo, Sweden
- University College London Hospital, London, United Kingdom

REFERENCES:
- [Background] Spencer R, Ambler G, Brodszki J, Diemert A, Figueras F, Gratacos E, Hansson SR, Hecher K, Huertas-Ceballos A, Marlow N, Marsal K, Morsing E, Peebles D, Rossi C, Sebire NJ, Timms JF, David AL; EVERREST Consortium. EVERREST prospective study: a 6-year prospective study to define the clinical and biological characteristics of pregnancies affected by severe early onset fetal growth restriction. BMC Pregnancy Childbirth. 2017 Jan 23;17(1):43. doi: 10.1186/s12884-017-1226-7. PMID 28114884
- [Derived] Bray G, Maksym K, Dilipkumar M, Spencer RN, Ginsberg Y, Weissbach T, Peebles DM, Marlow N, Huertas-Ceballos A, Buquis G, Okell J, Hecher K, Diemert A, Singer D, Hansson SR, Ley D, Figueras F, Gratacos E, Crispi F, David AL, Hunter R. Economic Impact of Severe Early-Onset Foetal Growth Restriction: A Multicentre Prospective Cohort Study. BJOG. 2026 Jan;133(1):61-70. doi: 10.1111/1471-0528.18266. Epub 2025 Jun 24. PMID 40552422
- [Derived] Spencer R, Maksym K, Hecher K, Marsal K, Figueras F, Ambler G, Whitwell H, Nene NR, Sebire NJ, Hansson SR, Diemert A, Brodszki J, Gratacos E, Ginsberg Y, Weissbach T, Peebles DM, Zachary I, Marlow N, Huertas-Ceballos A, David AL. Maternal PlGF and umbilical Dopplers predict pregnancy outcomes at diagnosis of early-onset fetal growth restriction. J Clin Invest. 2023 Sep 15;133(18):e169199. doi: 10.1172/JCI169199. PMID 37712421
- [Derived] Lingam I, Okell J, Maksym K, Spencer R, Peebles D, Buquis G, Ambler G, Morsing E, Ley D, Singer D, Tenorio V, Dyer J, Ginsberg Y, Weissbach T, Huertas-Ceballos A, Marlow N, David A; EVERREST consortium. Neonatal outcomes following early fetal growth restriction: a subgroup analysis of the EVERREST study. Arch Dis Child Fetal Neonatal Ed. 2023 Nov;108(6):599-606. doi: 10.1136/archdischild-2022-325285. Epub 2023 Apr 26. PMID 37185272